CLINICAL TRIAL: NCT03036696
Title: The Breastfeeding and Early Child Health (BEACH) Interview Study
Brief Title: The BEACH Interview Study- Pregnant and Breastfeeding Mothers
Acronym: BEACH
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601909
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Pediatric Obesity; Recruitment
Keywords: Retention; Lactation; Human milk; Pregnancy; Clinical Research Studies; BEACH
MeSH Terms: conditions — Pediatric Obesity; Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Non-invasive biospecimens include stool, saliva, blood, urine, human milk, and vaginal swab.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant Mothers Interview: (1) 18 years old or over, (2) between 28-38 weeks of pregnancy, (3) lives in Gainesville, Florida, and (4) are committed to exclusively breastfeeding through 6 months.
  Interventions: Other: Pregnant Mothers Interview
- Breastfeeding Mothers Interview: (1) 18 years old or over, (2) actively breastfeeding infant less than 12 months of age, and (3) lives in Gainesville, Florida.
  Interventions: Other: Breastfeeding Mothers Interview

INTERVENTIONS:
Other: Pregnant Mothers Interview — Pregnant mothers will be interviewed and asked to provide feedback on common strategies used for recruitment, challenges that would preclude them from enrolling and participating in CRTs, their preferences for incentives, data collection, bio-specimen collection and preferences for methods related to non-invasive sample collection.
  Data collection for pregnant mothers includes Clinical Health Update (3rd trimester) and Physical Activity questionnaires.
  The following will be collected from mothers during the interview: self-reported behavioral data, maternal human milk (HM), stool, urine, saliva, and vaginal swab.
  Groups: Pregnant Mothers Interview
Other: Breastfeeding Mothers Interview — Breastfeeding mothers will be interviewed and asked to provide feedback on common strategies used for recruitment, challenges that would preclude them from enrolling and participating in CRTs, their preferences for incentives, data collection, bio-specimen collection, and preferences for methods related to non-invasive sample collection.
  Data collection for breastfeeding mothers includes Clinical Health update (post-natal), Infant Feeding, and Physical Activity questionnaires.
  The following will be collected from mothers during the interview: self-reported behavioral data, maternal human milk (HM), stool, urine, saliva, and vaginal swab.
  Groups: Breastfeeding Mothers Interview

SUMMARY:
Interview pregnant and breastfeeding mothers in the Gainesville, FL area to optimize; clinical study recruitment and retention, patient-centered outcomes, and stool collection procedures.

DETAILED DESCRIPTION:
This is an interview study that will enroll mothers during 28 weeks or greater of pregnancy and assess recruitment, patient-centered outcomes, and stool collection procedures via individualized interviews and data collection. Participants will be recruited from the greater Gainesville, FL area. Data collection will include questionnaires/surveys as well as minimal risk non-invasive biological samples such as stool, human milk, saliva, vaginal swab, and urine collection. Participants will be seen at a location convenient for them.

ELIGIBILITY:
Inclusion Criteria:

* Females 18>45, between 28-38 weeks pregnant, lives in Gainesville, Florida, and committed to exclusively breastfeeding through 6 months.
* Females 18>45, actively breastfeeding for <12 months and lives in Gainesville, Florida

Exclusion Criteria:

* Mothers who do not plan to exclusively breastfeed their infant for at least the first 6 months or actively breastfeeding.
* Mothers who do not live in Gainesville, FL
* Mothers who are not between the ages of 18-45
* Mothers who are not between 28-38 weeks of gestation or a breastfeeding mother.
* Mothers who have only one breast which is capable of producing milk and/or have a history of inadequate milk production.
* Mothers who have consumed alcohol during this pregnancy.
* Mothers who have abused drugs during this pregnancy.
* Mothers who have smoked during this pregnancy.
* Mothers who have been diagnosed with pre-eclampsia during this pregnancy.
* Mothers who have had a previous pre-term delivery (baby born 2 months before the due date or <35 weeks).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The research team will recruit pregnant women (n = 30) and breastfeeding mothers' (n = 30) paired with infant (n=30) to participate in individual, in-depth, semi structured, and audio-recorded interviews.
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Strategies for recruiting and retaining pregnant and breastfeeding mothers into clinical research studies (CRTs) will be measured by way of interview. | 6 months
  Interviews will be analyzed to determine the efficacy of common strategies used to recruit pregnant and breastfeeding mothers into CRTs, challenges or barriers that would preclude women from enrolling and participating in CRTs, their preferences for incentives, as well their preference and methods related to non-invasive sample collection.

SECONDARY OUTCOMES:
Measure bioactive compounds in human milk (HM) via Enzyme-linked immunosorbent assay (ELISA) | 1 year
Quantify the infant intestinal gene expression profile in stool by real-time polymerase chain reaction (PCR) | 1 year
Measure the infant intestinal gene expression profile in stool via whole genome sequencing (WGS) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Lemas, PhD, Principal Investigator — University of Florida
Locations (1):
- Magda Francois, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH Data Sharing Policy of award 1U24DK097193, all data generated by Southeast Center for Integrated Metabolomics (SECIM), along with the corresponding metadata, will be deposited into the NIH Metabolomics Data Repository and Coordinating Center (DRCC) as soon as all quality control steps are completed. Data will be embargoed for one year and, after the expiration of the embargo, made visible to the scientific community regardless of publication status for the data.